CLINICAL TRIAL: NCT06126549
Title: A Randomized Trial to Compare Effectiveness of Two Interventions for Caregivers of Patients With Acquired Brain Injury
Brief Title: Comparison of Two Interventions for Caregivers of Patients With Acquired Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shepherd Center, Atlanta GA (Other)
Responsible Party: Principal Investigator, Michael Jones, Director Emeritus, Virginia C Crawford Research Institute, Shepherd Center, Atlanta GA
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 835
Record Dates: First submitted 2023-11-06; First posted 2023-11-13 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Acquired Brain Injury
Keywords: Acquired Brain Injury; Inpatient Rehabilitation; Family Caregivers; Caregiver Stress; Caregiver Self-Efficacy
MeSH Terms: conditions — Brain Injuries; Caregiver Burden

STUDY DESIGN:
Intervention Model Description: Evaluation of two interventions to usual care, comparing change over time in three outcome measures: caregiver stress, caregiver depression, caregiver perceived self-efficacy in care management
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care (Active Comparator): Usual Care (UC) consists of nurse instruction in care routines, case management family support for discharge, referral to family counseling and community services as indicated, and general information resources about brain injury. Usual Care participants also have access to peer support services, including peer mentoring, brain injury education classes, and workshops for caregivers.
  Interventions: Behavioral: Usual Care
- Building Better Caregivers (Active Comparator): Building Better Caregivers (BBC) was developed for caregivers of patients with Alzheimers' Disease and has been adapted for caregivers of patients with ABI. BBC is a peer-led, problem-solving intervention delivered in 6 group workshop sessions. Key components include problem-solving; making an action plan; managing stress and fatigue, difficult care partner behavior, and difficult thoughts/emotions. Each of the workshops last 60 minutes and usually take place once a week over a 6-8 week span of time.
  Interventions: Behavioral: Building Better Caregivers; Behavioral: Usual Care
- Problem Solving Training (Active Comparator): Problem Solving Training (PST) is a clinician-led intervention, administered one-on-one via phone calls, assigned readings, and practice assignments between calls. PST teaches caregivers how to address problems and apply a specific problem-solving technique that calls for brainstorming, consideration, development, and evaluation to address current problems the caregiver may be facing. The training aims to teach the strategy, so caregivers can apply it in the present, as well as the future. Each of the 6 Problem Solving Training Sessions last from 30-60 minutes and usually take place once a week over a 6-week span of time.
  Interventions: Behavioral: Problem Solving Training; Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Building Better Caregivers — Peer-led, group intervention for caregivers focused on problem-solving
  Arms: Building Better Caregivers
Behavioral: Problem Solving Training — Clinician-led, one-to-one intervention for caregivers focused on problem-solving
  Arms: Problem Solving Training
Behavioral: Usual Care — Usual discharge training and support offered to family caregivers of ABI patients

SUMMARY:
The goal of this clinical trial is to compare effectiveness of two interventions for family caregivers of patients with acquired brain injury who are transitioning home after inpatient rehabilitation. The main question it aims to answer is whether these interventions reduce caregiver stress and burden, compared to usual care. Secondary effects include the impact on caregivers' depressive symptoms and perceived self-efficacy as a caregiver. The study will also try to determine if caregivers will engage in these interventions during the acute (inpatient rehabilitation) stage of injury.

Participants in the study are family members of the ABI patient, aged 18 year or older, who will be responsible for the patient's care and supervision once discharged home from inpatient rehabilitation. The two interventions, one clinician-led and one peer-led, will be compared to usual care.

DETAILED DESCRIPTION:
This study will evaluate effectiveness of two problem-solving training interventions on caregivers' emotional health and well-being (stress, depressive symptoms, caregiving self-efficacy). Participants are family members of patients with acquired brain injuries (ABI) admitted for inpatient rehabilitation, with a planned discharge home. Caregivers who agree to participate will be randomly assigned to one of three family support interventions. The Building Better Caregiver program is a peer-led group intervention. Problem Solving Training is an individual clinician-led intervention. Both interventions aim to equip caregivers with problem solving tools. The third intervention is existing support and assistance for family members who will be caregivers for patients discharged home after inpatient rehabilitation. This Usual Care is available to all three groups and consists of nurse instruction in care routines, case management family support for discharge, referral to family counseling and community services as indicated, and general information resources about brain injury.

Caregiver-reported outcome measures (CROs) will be collected in three domains: 1) caregiver stress/burden and emotional health, 2) caregiver perceived self-efficacy in managing their loved-one's care needs, and 3) healthcare utilization by patient and caregiver. We will use three standardized outcome measures: 1) Kingston Caregiver Stress Scale (KCSS), 2) Patient Health Questionnaire (PHQ-9), and 3) Revised Scale for Caregiving Self-Efficacy (SCS-E). The measures will be collected at four timepoints: upon enrollment in the study ("Pre"), within 72 hours of discharge (D/C), and 30 and 90 days post-discharge. The impact of each intervention on the rate of patients' 30-day, unplanned hospital readmissions will also be examined.

ELIGIBILITY:
Inclusion Criteria:

* Family member of patients admitted to inpatient rehabilitation for acquired brain injury, with a planned discharge to home.
* Able to begin intervention before discharge
* Able to speak and understand English or Spanish

Exclusion Criteria:

* Patient's discharge location is not to home

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Kingston Caregiver Stress Scale (KCSS) | 1) baseline, at time of enrollment in the study and prior to randomization; 2) within 72 hours of discharge to home; 3) 30-days post-discharge; 90-days post-discharge
  Caregiver stress and burden; scores range from 10-50; higher score reflects higher stress

SECONDARY OUTCOMES:
Patient Health Questionnaire - 9 (PHQ-9) | 1) baseline, at time of enrollment in the study and prior to randomization; 2) within 72 hours of discharge to home; 3) 30-days post-discharge; 90-days post-discharge
  Caregiver depressive symptoms; scores range from 0-27; higher score reflects higher depression
Revised Scale for Caregiving Self-Efficacy (SCS-E). | 1) baseline, at time of enrollment in the study and prior to randomization; 2) within 72 hours of discharge to home; 3) 30-days post-discharge; 90-days post-discharge
  Contains 15 items within 3 subscales (self-efficacy for obtaining respite, responding to disruptive patient behaviors, and controlling upsetting thoughts about caregiving). Items are rated on a 0-100 scale.

OTHER OUTCOMES:
Patient unplanned hospital readmissions | Assessed by telephone follow-up interview 30-40 days post-discharge
  Hospital-wide assessment of number and duration of unplanned hospital readmissions in the 30 days post-discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Shepherd Center, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No